CLINICAL TRIAL: NCT05662046
Title: Deformity of the Forefoot in Children With Unilateral Cerebral Palsy
Acronym: Mediopied-PC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Mediopied-PC
Record Dates: First submitted 2019-03-28; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Forefoot Adductus; Cerebral Palsy
Keywords: Cerebral Palsy; Forefoot Deformity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Midfoot and backfoot deformities are well described in children with Cerebral palsy. However, data regarding forefoot deformities in Cerebral palsy remain scarce in a population were foot deformities are the most frequent musculo-skeletal deformities.

DETAILED DESCRIPTION:
Foot deformities are the most frequent musculo-skeletal deformities in children with Cerebral palsy. Pain starts in the foot, especially during gait in Cerebral Palsy Children (GMFCS I and II) and induce gait limitations, balance disorders, wounds, aesthetic disorders and difficulties to support shoes.

Metatarsus Adductus is the most common foot deformity in children with or without disorder, occuring on 1-2/1000 births. In 4 to 14% of the children, evolution is not favorable at 5 years. In that case, the diagnostic of Cerebral palsy have to be considered.

ELIGIBILITY:
Inclusion Criteria:

* Child who benefit a standardised clinical evaluation before a 3D Gait Analysis with forefoot deformity measure
* Child age less than 18 years old
* Child with left or right unilateral cerebral palsy
* Walking child ( GMFCS score I, II or III)
* In case of several 3D Gait Analysis for the child: the 3D gait analysis was chosen first before any local spasticity treatment with botulinic toxin injection or the 3D gait evaluation the more far from local spastica treatment with botulinic toxin injection was chosen in second .

Exclusion Criteria:

* Hemiplegia due to another etiology
* History of lower limb or foot surgery before the clinical evaluation
* Local spasticy treatment with botulinic toxin injection less than 3 months before the clinical evaluation
* Participation refusal

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Walking child with unilateral Cerebral Palsy who benefit of a 3D Motion Analysis on the motion analysis laboratory in Brest, France, between august 2012 and may 2017.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Measure of the forefoot deformity prevalence in plegia and non-plegia foot during gait in unilateral cerebral palsy children | 1 day
  we report in our population the forefoot axis measured by the angle between the heel bisector and the axis between the second and third metatarsal.

SECONDARY OUTCOMES:
Anthropometric factors (age) associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the age (years mean, standard deviation) of the patients CP
Anthropometric factors (sexe) associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the sexe of the patients (female or male)
Anthropometric factors (type of cerebral palsy)associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the plegia side of the patients cerebral palsy : right or left
functional factors associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the GMFCS score of the patients cerebral palsy : GMFCS 1, 2, 3, 4 or 5 (4-5 non ambulant 1-3 ambulant children)
biomechanical osteoarticular factors associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report biomechanical osteoarticular factors : hindfoot axis, foot dorsiflexion, footprint, tibial torsion, femoral antetorsion, leg length inequality) , Spasticity of lower limb muscle (Modified Ashworth Scale and Tardieu Scale) and Motricity of lower limb muscle ( Boyd scale and MRC evaluation)
Spasticity factors associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the Spasticity of lower limb muscle (Modified Ashworth Scale and Tardieu Scale)
Motricity factors associated with forefoot deformities on plegia side in walking children with unilateral Cerebral Palsy. | 1 day
  we report the motricity of lower limb muscle ( Boyd scale and MRC evaluation)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Houx, Brest
  - PRIGENT, Concarneau

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.